CLINICAL TRIAL: NCT01224392
Title: Randomized Trial of Preoperative Radiotherapy With an Integrated Simultaneous Boost Compared to Chemoradiotherapy for T3-4 Rectal Cancer
Brief Title: Simultaneous Integrated Boost Preoperative Radiotherapy for Rectum Cancer
Acronym: RectumSIB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Mark De Ridder, Head of Radiotherapy Department, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RectumSIB
Record Dates: First submitted 2010-06-28; First posted 2010-10-20 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Rectal Cancer
Keywords: colorectal cancer; colorectal neoplasms; radiotherapy; chemoradiotherapy; T3-4 rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms | interventions — Chemoradiotherapy; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concomitant chemoradiotherapy (Active Comparator): Radiotherapy (23 x 2 Gy) + capecitabine 825mg/m2 p.o. twice daily, excluding weekends
  Interventions: Other: Chemoradiotherapy
- Radiotherapy with boost (Experimental): Radiotherapy (23 x 2 Gy), with a simultaneous integrated boost up to 55.2 Gy on the primary tumor
  Interventions: Radiation: Radiotherapy with boost

INTERVENTIONS:
Other: Chemoradiotherapy — Radiotherapy (23 x 2 Gy) + capecitabine 825mg/m2 p.o. twice daily, excluding weekends
  Other Names: Xeloda (capecitabine)
  Arms: Concomitant chemoradiotherapy
Radiation: Radiotherapy with boost — Radiotherapy (23 x 2 Gy), with a simultaneous integrated boost up to 55.2 Gy on the primary tumor
  Other Names: Preoperative radiotherapy
  Arms: Radiotherapy with boost

SUMMARY:
The investigators propose a randomized non-inferiority trial that compares preoperative Fluoro Uracil (FU)-based chemoradiotherapy to radiotherapy with a simultaneous integrated boost. In patients with T3-4 rectal cancer, the latter approach is considered preferential with regard to toxicity and cost. The metabolic response of the tumor, as assessed by 18F-2-Fluoro-2-Deoxyglucose-Positron Emission tomography (18F-FDG PET) or PET-CT, will be used as a surrogate marker of cause specific outcome

ELIGIBILITY:
Inclusion Criteria:

* histopathologically confirmed rectal adenocarcinoma with an inferior border within 15 cm of the anal verge
* the tumor has to have evidence of T3 or T4 disease on Magnetic Resonance Imaging (MRI) or endoluminal ultrasound

Exclusion Criteria:

* unresectable metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status > 3
* patients not deemed fit for radiotherapy, capecitabine or surgery
* pregnant or lactating patients
* women with child bearing potential who lack effective contraception
* patients below 18 years old

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2010-01; Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
reduction in metabolic tumor activity | at baseline and at 5 to 6 weeks after neo-adjuvant therapy

SECONDARY OUTCOMES:
histological downgrading (Dworak classification) | after the rectum surgery
  pathological evaluation of surgical resection specimens
number of R0, R1 and R2 resections | after the rectum surgery
  pathological evaluation of surgical resection specimens
acute and late toxicity, according to the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events v3.0 (CTCAE) | at baseline, every 6 months after completion of radiotherapy and then yearly until 3 years
local control | every 6 months in the first year after completion of radiotherapy and then yearly until 3 years
progression free survival | every 6 months in the first year after completion of radiotherapy and then yearly until 3 years
survival | every 6 months in the first year after completion of radiotherapy and then yearly until 3 years
  overall survival
quality of life | at baseline, every 6 months in the first year after completion of radiotherapy and then yearly until 3 years
cost evaluation | during the treatment and follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Mark De Ridder, Prof.Dr., Principal Investigator — UZ Brussel, Vrije Universiteit Brussel, dienst Radiotherapie
Locations (2):
- Belgium (2):
  - UZ Brussel , Vrije Universiteit Brussel, dienst Radiotherapie, Jette, Brussels Capital
  - UZ Brussel, Vrije Universiteit Brussel, dienst Radiotherapie, Jette